CLINICAL TRIAL: NCT05902312
Title: Comparative Effectiveness of Repetitive Versus Deep Transcranial Magnetic Stimulation for Major Depression: A Randomized Controlled Trial
Brief Title: Repetitive Versus Deep Transcranial Magnetic Stimulation for Major Depression
Acronym: ReDeeMD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-11389
Record Dates: First submitted 2023-05-31; First posted 2023-06-13 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
Keywords: MDD; TMS; deep TMS
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: randomized, single-center, two-arm, parallel-group superiority trial
Who Masked: Outcomes Assessor
Masking Description: Given the study's design, blinding participants and TMS operators will not be possible. Still, staff responsible for participant assessments and data analysis will be blinded to treatment conditions and external to the clinic staff. Patients will be instructed not to reveal their group assignment to the raters. Patients will not be given the specifics of the treatment parameters and will be instructed not to talk to each other during the study period. Both treatments will be presented as effective to them. Lastly, the data management center will strictly control access to the randomization code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- repetitive Transcranial Magnetic Stimulation (Active Comparator): rTMS on a MagPro X100 research grade stimulator (MagVenture) equipped with a B70 fluid-cooled coil. Participant will receive the MDD FDA-approved iTBS protocol (triplet 50 Hz bursts repeated at 5 Hz, 2 s ON and 8 s OFF; 600 pulses per session; total duration of 3 min 9 s, 120% hand motor threshold)
  Interventions: Device: transcranial magnetic stimulation
- deep Transcranial Magnetic Stimulation (Experimental): dTMS on a research Brainsway system equipped with an H7-Coil. Participants will receive the MDD FDA-cleared 18 Hz stimulation protocol (2 sec ON, 20 sec OFF, 55 trains; 1980 pulses per session; 20 min 10 s duration; 120% hand motor threshold)
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — Participants will receive either rTMS or dTMS
  Other Names: deep transcranial magnetic stimulation

SUMMARY:
The goal of this randomized controlled trial is to he effectiveness of two different TMS techniques in TRD, repetitive TMS (rTMS) and deep TMS (dTMS). The main questions it aims to answer are:

type of study: clinical trial participant population/health conditions : Major Depressive Disorder To assess the superiority of dTMS over rTMS in TRD To evaluate the predictive capacity of scalable candidate biomarkers Participants will be randomly allocated to one of the two intervention groups (rTMS or dTMS).

DETAILED DESCRIPTION:
The primary aim of this trial is to compare the effectiveness of two different TMS techniques in TRD, repetitive TMS (rTMS) and deep TMS (dTMS). Compared to rTMS, dTMS delivers a broader magnetic field, which in turn reduces coil positioning error and maximizes the probability of optimal cortical stimulation. A past RCT comparing both approaches found a greater depression score decrease and response/remission rates for dTMS, but was short of reaching significance for remission rates (primary outcome). Critical components of this RCT were suboptimal, including too few treatment sessions and insufficient statistical power, both of which could have obscured an actual difference between modalities. Proof of a more effective type of TMS over another would translate into increased odds of improvement for TRD patients who live with a chronic and disabling illness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Major Depressive Disorder, at least moderate intensity, single or recurrent episode
* HRSD-17 score of at least 18
* No improvement to at least two adequate courses of antidepressants (based on the ATHF) or were unable to tolerate at least two separate trials of antidepressants of inadequate dose and duration
* On a stable antidepressant regimen for the past four weeks before screening
* Patients with a chronic depressive episode >2 years and who have previously received ECT or ketamine will be eligible to participate

Exclusion Criteria:

* Having previously received TMS;
* Substance use disorder within the last three months
* Diagnosis of bipolar or psychosis spectrum disorder
* Anxiety or personality disorder that is assessed by a study investigator to be the primary cause and causing greater impairment than MDD
* Concomitant major unstable medical or neurological illness
* Intracranial implant, cardiac pacemaker or implanted medication pump
* Significant laboratory abnormality;
* Active suicidal intent
* Pregnancy
* If participating in psychotherapy, must have been in stable treatment for at least three months before entry into the study, with no anticipation of change
* Currently taking more than the equivalent of 2 mg of lorazepam of a benzodiazepine daily or any dose of an anticonvulsant due to the potential to limit TMS effectiveness

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression-17 (HRSD-17) | Baseline to Week 6
  score change. Higher score means worse outcome. (Min = 0, Max = 53)
Response (yes/no) on Hamilton Rating Scale for Depression-17 | baseline to Week 6
  Defined as a score reduction of 50% or more
Remission (yes/no) on Hamilton Rating Scale for Depression-17 | Week 6
  Defined as a score of 7 or less

SECONDARY OUTCOMES:
Hamilton Rating Scale for Depression-17 | Baseline to Week 7
  score change. Higher score means worse outcome. (Min = 0, Max = 53)
Hamilton Rating Scale for Depression-17 | Baseline to Week 10
  score change. Higher score means worse outcome. (Min = 0, Max = 53)
Hamilton Rating Scale for Depression-17 | Baseline to Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 53)
Response (yes/no) on Hamilton Rating Scale for Depression-17 | Baseline to Week 7
  Defined as a score reduction of 50% or more
Response (yes/no) on Hamilton Rating Scale for Depression-17 | Baseline to Week 10
  Defined as a score reduction of 50% or more
Response (yes/no) on Hamilton Rating Scale for Depression-17 | Baseline to Week 18
  Defined as a score reduction of 50% or more
Remission (yes/no) on Hamilton Rating Scale for Depression-17 | Baseline to Week 7
  Defined as a score of 7 or less
Remission (yes/no) on Hamilton Rating Scale for Depression-17 | Baseline to Week 10
  Defined as a score of 7 or less
Remission (yes/no) on Hamilton Rating Scale for Depression-17 | Baseline to Week 18
  Defined as a score of 7 or less
Hamilton Rating Scale for Depression-28 | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 90)
Hamilton Anxiety Rating Scale (HAM-A) | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 56)
Quick Inventory of Depressive Symptomatology (self-report) (QIDS-SR 16) | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 42)
General Anxiety Disorder-7 (GAD-7) | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 21)
Snaith-Hamilton Pleasure Scale (SHAPS) | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min= 0, Max = 56)
Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 30)
Rumination Response Scale (RRS) | Baseline to Week 6, Week 7, Week 10, Week 18
  score change. Higher score means worse outcome. (Min = 0, Max = 88)
Adult AHDH Self-Report Scale | Baseline to Week 18
  qualitative.
McLean Screening Instrument for Borderline Personality Disorder | Baseline
  score. Higher score means worse outcome. (Min = 0, Max = 10)
World Health Organization Quality of Life Short Version (WHOQOL-BREF) | Baseline to Week 6, Week 7, Week 10, Week 18
  Difference score. Lower score means worse outcome. (Min = 26, Max = 130)
Cognitive Difficulties Scale (MacNair-R) | Baseline to Week 6, Week 7, Week 10, Week 18
  Difference score. Higher score means worse outcome. (Min = 0, Max = 156)
Memory Complaints Scale (MacNair) | Baseline to Week 6, Week 7, Week 10, Week 18
  score. Higher score means worse outcome. (Min = 0, Max = 45)
Visual Pain Scale | Each treatment day
  Maximum score (during treatment). Higher score means worse outcome. (Min = 0, Max = 10).
Sex and Gender scale | Baseline
  Descriptive statistics

OTHER OUTCOMES:
Electroencephalogram to predict treatment response | Baseline
  individual alpha frequency
Electroencephalogram event-related potentials | Baseline
  Reward positivity
Electrocardiogram | Baseline
  corrected QT interval
Pupil measures | Baseline
  pupil reactivity measures

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Miron, MD PhD, Principal Investigator — Centre de Recherche du Centre Hospitalier de l'Université de Montréal
Locations (1):
- CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-26): https://cdn.clinicaltrials.gov/large-docs/12/NCT05902312/Prot_SAP_000.pdf